CLINICAL TRIAL: NCT00138073
Title: Effectiveness of a Web-Based Computer Application in Improving Pulmonary Artery Catheter Waveform Interpretation Among Nurses and Physicians
Brief Title: Effectiveness of a Computer Application in Improving Pulmonary Artery Catheter Waveform Interpretation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of lack of resources to complete it.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jaime Chang, MD, Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2005-P-001381/1; MGH
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Artery Catheter Waveform Interpretation
Keywords: pulmonary artery catheter; waveform interpretation; computer-based learning; medical education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Web-based waveform interpretation guide (Experimental): The arm has access to the Web-based waveform interpretation guide.
  Interventions: Device: Web-based waveform interpretation guide

INTERVENTIONS:
Device: Web-based waveform interpretation guide — Use of an educational website.

SUMMARY:
Skill with pulmonary artery catheter (PAC) waveform interpretation is inadequate among physicians and nurses. We, the investigators at Massachusetts General Hospital, have developed a web-based computer program to assist physicians and nurses in PAC waveform interpretation. We will study the effectiveness of this program on improving the interpretation of waveforms on a computer-based test.

DETAILED DESCRIPTION:
The pulmonary artery catheter (PAC) guides diagnosis and treatment in the intensive care unit (ICU), but studies have shown that physicians and nurses collectively have inadequate skill in interpreting PAC waveforms. We have developed a Web-based application that provides physicians and nurses with rapid access to relevant PAC-related content for use in patient care situations. The application begins with a visual index that assists clinicians in the recognition of both normal and abnormal waveforms and provides waveform-specific links to concise advice on making accurate pressure measurements, troubleshooting system problems, and avoiding complications of catheter use. Initial evaluation will consist of a before-and-after trial to determine whether the application improves test performance in the areas of waveform recognition, accuracy of measurement, and appropriateness of action. Once the resource is in production, we will electronically log usage and survey users to evaluate the extent and effect of actual utilization.

ELIGIBILITY:
Inclusion Criteria:

* Critical care nurses
* House officers rotating through the medical Intensive Care Unit
* Fellows rotating through the medical Intensive Care Unit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Octo Barnett, MD, Principal Investigator — Massachusetts General Hospital/Laboratory of Computer Science
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Web-based Waveform Interpretation Guide
Started | 55
Pre-intervention Testing | 55
Completed | 0
Not Completed | 55
Not completed — lack of resources | 55

BASELINE CHARACTERISTICS:
Arm/Group | Web-based Waveform Interpretation Guide
Number analyzed (Participants) | 55
Age, Customized [Number; unit: participants] — Baseline measure of age was not collected.
  participants
    any age | 55
Sex/Gender, Customized [Number; unit: participants] — Baseline measure of gender was not collected.
  participants
    any gender | 55
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Score on a Computer-based Test on Pulmonary Artery Catheter Waveform Interpretation
Description: The study was terminated before the primary outcome could be measured. None of the participants took the post-intervention test.
Time Frame: 1 month
Arm/Group | Web-based Waveform Interpretation Guide
Number analyzed (Participants) | 0

2. Secondary Outcome: Individual and Collective Frequency of Use and Usage Patterns of the Web-based Waveform Interpretation Guide
Description: The study was terminated before the secondary outcome could be measured. Usage data was not collected over the following year.
Time Frame: 1 year
Arm/Group | Web-based Waveform Interpretation Guide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: The participants had access to instructional information on a website. No adverse events were expected therefore none were collected.
Arm/Group | Web-based Waveform Interpretation Guide
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes